CLINICAL TRIAL: NCT02461394
Title: User Performance Evaluation of Contour Plus, Accu-Chek Active, Accu-Chek Performa and OneTouch Select Simple Blood Glucose Monitoring Systems Following ISO 15197:2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1469-BL
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

INTERVENTIONS:
Device: Blood glucose monitoring systems for self-testing
  Other Names: Contour Plus, Accu-Chek Active, Accu-Chek Performa, OneTouch Select Simple

SUMMARY:
The user performance evaluation shows whether people with diabetes are able to obtain accurate measurement results with a blood glucose monitoring system. In this study, user performance evaluation will be performed for Contour Plus (Bayer Healthcare Diabetes Care), Accu-Chek Active (Roche Diagnostics), Accu-Chek Performa (Roche Diagnostics) and OneTouch Select Simple (LifeScan) following ISO 15197:2013, clause 8.

The study will be performed in 2 parts. Each part will comprise testing of 2 BGMS.

For each BGMS, measurement procedures for user performance evaluation will be performed with 1 test meter and 1 reagent system lot by the study subjects.

The same meter and an additional test meter will be used for double measurements performed by study personnel (with the same reagent system lot used by subjects).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or no diabetes
* For provoked blood glucose excursions due to insulin dose adjustment: Male or female with type 1 diabetes or type 2 diabetes and intensified insulin therapy or insulin pump therapy.
* Minimum age of 18 years
* Signed informed consent form
* Legally competent and capable to understand character, meaning and consequences of the study

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Physical or mental constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Incapability of giving informed consent
* < 18 years
* Legally incompetent
* Accommodated in an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent from investigator or sponsor
* For provoked blood glucose excursions 50 - 80 mg/dl:
* Coronary heart disease
* Condition after myocardial infarction
* Cerebral incidence
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Acceptance criteria defined by ISO 15197:2013 (see description) | For each subject, the experimental phase has an expected duration of up to 3 hours
  95 % of the individual glucose measured values shall fall within ± 15 mg/dl (0.83 mmol/l) of the measured values of the comparison measurement procedure at glucose concentrations < 100 mg/dl (5.55 mmol/l) and within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany